CLINICAL TRIAL: NCT05773287
Title: Targeted Health Coaching Intervention to Improve Physical Activity Maintenance and Mobility Post-Structured Cardiac Rehabilitation Programming Among Older Adults: A Pilot Study
Brief Title: Targeted Health Coaching to Improve Physical Activity Post-Structured Cardiac Rehabilitation
Acronym: Target-CR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00112929; 1P30AG064201-01 (NIH)
Record Dates: First submitted 2023-03-10; First posted 2023-03-17 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Rehabilitation; Health Coaching; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Health Coaching Group (Experimental)
  Interventions: Behavioral: Targeted Health Coaching Group
- Standard Care Group (Placebo Comparator)
  Interventions: Behavioral: Standard Care Group

INTERVENTIONS:
Behavioral: Targeted Health Coaching Group — Participants in the THC group will receive an exercise prescription (steps/day) based on their last cardiac rehabilitation session exercise prescription. Participants will be provided a Garmin wearable device to track steps/day. Additionally, participants will partake in 6 virtual or in-person health coaching sessions lasting approximately 30-60 minutes in duration. These sessions will take place approximately every other week during the 3-month intervention period.
  Arms: Targeted Health Coaching Group
Behavioral: Standard Care Group — Participants in the SC group will receive an exercise prescription (steps/day) based on their last cardiac rehabilitation session exercise prescription. Participants will be provided a Garmin wearable device to track steps/day. Additionally, participants will be provided with a single virtual or in-person education session, lasting approximately 30 minutes, at the beginning of the 3-month intervention period.
  Arms: Standard Care Group

SUMMARY:
To identify factors and triggers influencing physical activity (PA) participation after structured cardiac rehabilitation (CR) among older adults who have enrolled in a center-based CR program, and compare the effects of a targeted health coaching intervention versus standard care immediately following structured CR on PA maintenance and functional fitness.

DETAILED DESCRIPTION:
Approximately 800,000 individuals in the United States have a heart attack every year, with almost 1 in 4 of those individuals already having suffered a previous heart attack. Attending cardiac rehabilitation (CR) following a cardiovascular event improves cardiorespiratory fitness and health-related quality of life, as well as decreases the risk of future illness and death from heart disease. Unfortunately, once an individual finishes a CR program, continued participation in physical activity (PA) too often reverts to previous sedentary patterns, limiting beneficial health effects. Continued participation in PA post-CR is especially challenging among older adults - likely due to a lack of self-efficacy and confidence in their ability to perform PA due to either their age or other health conditions that make PA more challenging. However, the need to address other health conditions, in conjunction with the benefits of improved strength and mobility, makes continued PA participation following a structured CR program even more useful for older adults. Although individuals typically understand habitual participation in PA is good for their health, we poorly understand why some individuals successfully adhere to and maintain PA habits, while others succumb to barriers preventing them from maintaining the health benefits beyond CR. In addition to understanding factors and triggers influencing PA maintenance beyond CR, little research has developed or investigated interventions targeting this important transition period following structured CR programming to promote continued PA participation "at home". Therefore, this proposal aims to 1) identify factors and triggers influencing PA participation after a traditional 36-session CR program (Stage 0); and 2) test a targeted health coaching intervention using these identified triggers to optimize PA maintenance and mobility among older adults who completed a center-based CR program.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide informed consent to participate in the Target-CR Study
* Must be able to read and speak English well enough to provide informed consent and understand instructions
* Age ≥60 years
* Diagnosed with coronary heart disease
* Of adequate clinical stability to allow study participation
* Own a smartphone device for application download

Exclusion Criteria:

* Planned relocation during the 3-month study period
* Medical procedure scheduled within the 3-month study period that may limit physical activity (i.e., joint replacement)
* Decompensated heart failure
* Heart failure - New York Heart Association class IV
* Severe pulmonary hypertension
* End-stage renal disease
* Cardiac transplantation
* Impairment from stroke, injury, or other medical condition that would prevent participation in the intervention
* Dementia that would prevent participation in the intervention and following study protocols
* Any other illnesses that, in the opinion of the local clinician, would negatively impact or mitigate participation in and completion of the protocol
* Psychiatric illness (self-report and screening)

  * Hospitalization for any psychiatric condition within one year (self-report)
  * Integrative Health Coaching Mental Health Screening Questionnaire score >4 (screening)
* Participation in an inpatient substance abuse rehabilitation program within one year

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E. Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center For Living, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research is a Stage 0 and I pilot project that will involve a small sample (26 participants) in order to understand factors and triggers influencing physical activity participation immediately following a structured cardiac rehabilitation program and testing a targeted intervention approach to maintaining physical activity participation among older adults. Given the primary focus of this study will be intervention development and feasibility, we do not anticipate that sharing data will be of significant scientific or clinical merit. Therefore, we are not planning to share the data broadly. However, the structure of how we collect data, what data we collect, and how it will be monitored is part of the implementation and evaluation plan. Those materials will be made available.
Supporting Information: Study Protocol
Time Frame: No later than 1 year following completion of the funded project period.
Access Criteria: The project PI and Co-investigators who use the data will be made aware of the location of the data on the Duke University secure server. All other researchers will be asked to contact the project PI to discuss the secondary use of the data or the need for direct access beyond what will be made available on clinical trials.gov. All potential users will need to oblige to make no attempt to identify participants from de-identified data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care/Education Group: Standard Care Group: Participants in the SC group will receive an exercise prescription (steps/day) based on their last cardiac rehabilitation session exercise prescription. Participants will be provided a Garmin wearable device to track steps/day. Additionally, participants will be provided with a single virtual or in-person education session, lasting approximately 30 minutes, at the beginning of the 3-month intervention period.
Period: Overall Study
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (6.3) | 72.5 (8.0) | 70.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity as Measured by Steps Per Day
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
Number analyzed (Participants) | 7 | 6
steps per day | 1194 (1641) | 554 (1762)
Statistical Analysis 1: Comparison: Targeted Health Coaching Group vs Standard Care/Education Group; Test type: Superiority; p = 0.509, t-test, 2 sided — The a priori threshold for statistical significance was 0.05

2. Primary Outcome: Average Adherence to Physical Activity Prescription
Description: A metric of adherence to the steps/day prescription, calculated as (steps/day completed) divided by (steps/day prescribed) times 100 and averaged across the study period. Reported as the average adherence (percent) to the steps per day prescription across the three-month study period.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
Number analyzed (Participants) | 7 | 6
percent | 110.4 (26.8) | 102.7 (18.1)
Statistical Analysis 1: Comparison: Targeted Health Coaching Group vs Standard Care/Education Group; Test type: Superiority; p = 0.552, t-test, 2 sided — The a priori threshold for statistical significance was 0.05

3. Secondary Outcome: Change in Senior Fitness Test Score (SFT) - Chair Stands
Description: The chair stand test is similar to a squat test to measure leg strength, in which participants stand up repeatedly from a chair for 30 seconds. Reported as the number of completed chair stands in 30 seconds.
Time Frame: Baseline, 3 months
Population: One participant opted out of the post-intervention SFT due to medical issues.
Measure: Mean (Standard Deviation); unit: chair stands/30 seconds
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
Number analyzed (Participants) | 7 | 5
chair stands/30 seconds | 1.6 (3.1) | 2.2 (1.1)

4. Secondary Outcome: Change in Senior Fitness Test Score (SFT) - Arm Curls
Description: The Arm Curl test is a test of upper body strength and involves performing as many arm curls as possible in 30 seconds, while sitting in a chair. Reported as change in the number of arm curls completed in 30 seconds.
Time Frame: Baseline, 3 months
Population: One participant opted out of the post-intervention SFT due to medical issues.
Measure: Mean (Standard Deviation); unit: arm curls/30 seconds
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
Number analyzed (Participants) | 7 | 5
arm curls/30 seconds | 1.4 (1.5) | 2.8 (2.5)

5. Secondary Outcome: Change in Senior Fitness Test Score (SFT) - 6-minute Walk Test (6MWT)
Description: The 6MWT is reported as the distance walked in 6 minutes to the nearest meter.
Time Frame: Baseline, 3 months
Population: One participant opted out of the post-intervention SFT due to medical issues.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
Number analyzed (Participants) | 7 | 5
meters | 5.7 (9.4) | 3.6 (3.1)

6. Secondary Outcome: Change in Senior Fitness Test Score (SFT) - 2-Minute Step Test
Description: The 2-Minute Step Test is a measure of endurance or physical stamina, reported as change in the number of steps, marching in place, achieved in 2 minutes.
Time Frame: Baseline, 3 months
Population: One participant opted out of the post-intervention SFT due to medical issues.
Measure: Mean (Standard Deviation); unit: steps per 2 minutes
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
Number analyzed (Participants) | 7 | 5
steps per 2 minutes | 5.7 (9.4) | 3.6 (3.1)

7. Secondary Outcome: Change in Senior Fitness Test Score (SFT) - Sit & Reach
Description: The Sit & Reach test measures lower body flexibility, specifically hamstring flexibility. Reported as the change in distance reached in inches.
Time Frame: Baseline, 3 months
Population: One participant opted out of the post-intervention SFT due to medical issues.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
Number analyzed (Participants) | 7 | 5
inches | 0.9 (2.4) | 2.0 (7.3)

8. Secondary Outcome: Change in Senior Fitness Test Score (SFT) - Back Scratch Test
Description: The Back Scratch Test is a measure of upper body flexibility. This is reported as the change in distance between fingertip of the middle fingers on each hand in inches.
Time Frame: Baseline, 3 months
Population: One participant opted out of the post-intervention SFT due to medical issues.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
Number analyzed (Participants) | 7 | 5
inches | -0.1 (1.0) | 0.2 (1.3)

9. Secondary Outcome: Change in Senior Fitness Test Score (SFT) - Timed Up and Go Test
Description: The Timed Up and Go test measures speed, agility, and balance. This is reported as the average change in time to the nearest second among two trials.
Time Frame: Baseline, 3 months
Population: One participant opted out of the post-intervention SFT due to medical issues.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
Number analyzed (Participants) | 7 | 5
seconds | 0.03 (0.60) | 0.20 (0.60)

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Targeted Health Coaching Group | Standard Care/Education Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 1/7 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted Health Coaching Group (N=7) | Standard Care/Education Group (N=6)
Atrial Flutter (Cardiac disorders) | 0 | 1
Atrial Fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Nonsustained Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT05773287/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT05773287/ICF_000.pdf